CLINICAL TRIAL: NCT03420144
Title: Growth Hormone Therapy and Its Effect on Nitrogen Metabolism and Malnutrition in Liver Cirrhosis
Brief Title: Growth Hormone Therapy in Liver Cirrhosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr.Virendra Singh, Professor of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GH in cirrhosis
Record Dates: First submitted 2018-01-11; First posted 2018-02-05 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Cirrhosis, Liver
Keywords: Growth hormone; cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis | interventions — Growth Hormone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Medical Therapy (Active Comparator): Standard medical therapy: diuretics, lactulose, rifaximin, diuretics, albumin infusion, nutritional support (as required)
  Interventions: Drug: Standard Medical Therapy
- Growth hormone (Active Comparator): Growth Hormone: GH therapy is initiated at a low dose of 1U/day and titrated slowly upward to a maximum dose of 3U/day (based on IGF-1 levels) subcutaneously for 1 year.
  Interventions: Drug: Standard Medical Therapy; Drug: Growth Hormone

INTERVENTIONS:
Drug: Standard Medical Therapy — Standard Medical Therapy will include nutritional support, rifaximin, lactulose, bowel wash, albumin, diuretics, multivitamins and antibiotics as required
Drug: Growth Hormone — GH therapy is initiated at a low dose of 1U/day and titrated slowly upward to a maximum dose of 3U/day (depending on IGF-1 levels) subcutaneously for 1 year.
  Arms: Growth hormone

SUMMARY:
Liver cirrhosis (LC) is a leading cause of morbidity and mortality worldwide. Life- threatening complications of liver cirrhosis are ascites, gastrointestinal bleeding, variceal bleed, hepatic encephalopathy and hepatocellular carcinoma (HCC) which are associated with poor prognosis.The leading causes of liver cirrhosis include excess alcohol consumption, viral hepatitis and non-alcoholic fatty liver disease. Malnutrition is common in end-stage liver disease (cirrhosis) and is often associated with a poor prognosis. It occurs in all forms of cirrhosis with different etiology and prevalence ranges from 65 to 100% depending upon the methods used for nutritional assessment and the severity of liver disease. Nutritional state influences survival in patients with decompensated cirrhosis. Protein malnutrition manifested by reduced skeletal muscle mass and hypoalbuminemia, exist in patients with cirrhosis despite apparent adequate food consumption and these patients have a higher rate of complications and, overall, an increased mortality rate. Also, Malnutrition has significant implications for liver transplantation; patients with poor nutritional status before transplantation have increased complications and higher mortality rates postoperatively. Screening all patients with chronic liver disease for nutritional abnormalities can identify those at risk of developing preventable complications.

Malnutrition is commonly associated with protein catabolism and the protein catabolic state of cirrhosis is associated with severe growth hormone (GH) resistance, with low levels of insulin-like growth factor (IGF)-I and its major binding protein (IGFBP)-3.

GH therapy in cirrhosis has been shown to improve nitrogen economy and to improve the GH resistance in a small pilot study by Donaghy et al. Also, GH therapy of short duration has shown to increase IGF1 levels, IGFBP-3 levels in patients of cirrhosis. GH therapy has also shown to improve liver regeneration and protein synthesis after hepatectomy in patients of HCC with cirrhosis.

However there is scarcity of data on clinical impact of long term administration of GH therapy in patients of cirrhosis. Hence, we undertook the present study to study the effect of growth hormone on nitrogen economy, malnutrition and liver regeneration in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Decompensated Cirrhosis of liver irrespective of etiology

Exclusion Criteria:

* Acute on chronic liver failure (fulfilling either APASL or CANONIC criteria of ACLF)
* Splenic diameter of more than 18 cm
* Concomitant HCC or other active malignancy
* Upper gastrointestinal bleeding in the previous 7 days
* Portal vein thrombosis
* Severe renal dysfunction as defined by creatnine > 1.5mg/dl
* Severe cardiac dysfunction
* Uncontrolled diabetes (Hb A 1c ≥ 9) or diabetic retinopathy
* Acute infection or disseminate intravascular coagulation
* Active alcohol abuse in last 3 months
* Known hypersensitivity to GH
* HIV co-infection
* Pregnancy
* Refusal to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Improvement in Nutritional status based on CT L3 SMI score. | One year
  Nutritional status will be assesses by skeletal muscle index measurement using CT scan measurements at L3 level

SECONDARY OUTCOMES:
Improvement in BMI | One Year
Improvement in Mid arm muscle circumference(MAMC) | One year
Improvement in hand grip strength | One year
  Hand grip strength will be measured with the hydraulic hand dyanamometer in Kg/force.
Clinical improvement in liver function | One Year
  Occurrence of decompensations namely ascites, hepatic encephalopathy and variceal bleed
Biochemical improvement in liver function | One year
  Improvment in MELD score
Improvement in Quality of life | One Year
  Quality of life will be assessed using SF-36V2 Health Survey questionnaire
Improvement in liver regeneration | One Year
  By measuring hepatic parenchymal cell specific marker (CD 133) and cell proliferation marker (Ki-67) by immunohistochemistry.

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kumari S, De A, Kalra N, Singh V. Growth Hormone Therapy in Decompensated Cirrhosis: An Open-Label, Randomized Control Trial. Am J Gastroenterol. 2024 Jan 1;119(1):116-126. doi: 10.14309/ajg.0000000000002300. Epub 2023 Apr 27. PMID 37115908